CLINICAL TRIAL: NCT04504123
Title: MMP-9 Inhibition for Recalcitrant Wet Age-Related Macular Degeneration (AMD)
Brief Title: MMP-9 Inhibition for Recalcitrant Wet AMD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Elliott Sohn, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202001041
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Exudative Macular Degeneration; Wet Age-related Macular Degeneration
Keywords: Active choroidal neovascularization (CNV)
MeSH Terms: conditions — Wet Macular Degeneration | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: Doxycycline Hyclate 50 mg versus placebo capsule
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Over encapsulation with opaque purple capsule
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Doxycycline (Experimental): Participants received doxycycline hyclate 50 mg capsule orally once a day for 6 months
  Interventions: Drug: Doxycycline Hyclate
- Placebo (Placebo Comparator): Participants received placebo (inactive) capsule orally once a day for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline Hyclate — Doxycycline Hyclate capsules, USP 50 mg
  Other Names: Antibiotic - tetracycline compound
  Arms: Doxycycline
Drug: Placebo — Placebo
  Other Names: Inactive substance
  Arms: Placebo

SUMMARY:
Wet (or neovascular) form of age-related macular degeneration (wAMD) is the most common cause of blindness in the Western world. Currently, anti-vascular endothelial growth factor (VEGF) intravitreal injections (IVI) remain the standard-of-care treatment for wAMD. Previous studies show that about 90% of treated patients lose minimal visual function after 2 years of follow-up. There is still, a subset of 15% patients, incomplete responders, that do not improve and possibly worsen due to the persistence of sub-retinal fluid (with or without intra-retinal fluid) with chronic treatment.

The investigators plan to evaluate the effect of oral doxycycline versus placebo on the anatomic and functional outcomes in persistent sub-retinal eye fluid in neovascular wet age-related macular degeneration. This subset are incomplete or non-responders to current anti-VEGF intravitreal therapy.

DETAILED DESCRIPTION:
The investigators plan to conduct a double masked, randomized study to assess the effect of low dose, oral doxycycline 50 mg once a day versus placebo in patients with wet age-related macular degeneration who are incomplete responders to anti-VEGF extended treatment regimens.

The study will be conducted over 9 months with every 3 month assessments; 6 months administration period of doxycycline versus placebo (double masked, randomized) and a 3 month follow up period. The participant visits will occur during clinic visits for standard-of-care intravitreal injections (IVI).

Medical information will be acquired from the standard of care optical coherence tomography (OCT), visual acuity (VA), and IVI administered (number, frequency and type of drug).

Blood plasma and aqueous fluid (anterior chamber tap) samples and study drug tolerability will be obtained at baseline, 6 months and 9 months. Plasma will be obtained to assay for inflammatory markers: MMP-9 levels and questionnaires will be obtained on 1) vision quality of life, and 2) study drug tolerance at Baseline, 6 months and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Wet age-related macular degeneration (wAMD);
* Solely treated with anti-VEGF IVI for active CNV due to wAMD. However, enrolled patients can have other retinal pathologies such as diabetic retinopathy or vein occlusion for which they are not being treated with anti-VEGF IVI;
* Must have persistent sub-retinal with or without intra-retinal fluid due to active CNV from wAMD despite receiving at least three consecutive injections with any anti-VEGF agent;
* Must not have encountered previous side effects from tetracycline medications.

Exclusion Criteria - Ocular:

* History of uveitis (including endophthalmitis) or presence of intraocular inflammation;
* Presence of significant epiretinal membrane or macular hole causing distortion of macular anatomy;
* Presence of media opacity preventing discerning of fluid on OCT;
* Any prior ophthalmic surgery (including YAG or retinal laser) within the previous 3 months or anticipated need for any ophthalmic surgery (including cataract extraction) for 9 months following randomization;
* History of peribulbar corticosteroid injection to the studied eye or the fellow eye within the past 6 months;
* History of intravitreal triamcinolone acetonide injection to the studied eye within the past 4 months;
* An ocular condition (other than AMD) is present in the studied eye that, in the opinion of the investigator, might alter visual acuity during the course of the study (e.g., retinal vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, and Irvine-Gass syndrome);
* CNV due to causes other than wAMD;
* Inability to follow up at the 6th and 9th months time points after recruitment;
* Missing two or more consecutive injections during the six months treatment period;
* Patient requiring imminent need for IVI anti-VEGF medication switch or another treatment intervention, such as photodynamic therapy, during the 9 months trial period;
* Presence of fluid associated with geographic atrophy or disciform scar;
* Any patient with sub-retinal and/or intra-retinal fluid that is not due to CNV (eg, overlying areas of geographic atrophy;
* Any patient actively being actively treated for Irvine-Gass Syndrome.

Exclusion Criteria - Systemic:

* Patient with and/or who developed an unstable medical status (e.g., glycemic control, blood pressure, cardiovascular disease, individuals who are unlikely or unable to complete the 9 months trial period) in the opinion of the investigator;
* Significant renal disease (defined as a serum creatinine >2.5 mg/dL);
* Systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg;
* History of headaches associated with tetracycline therapy
* History of pseudotumor cerebri;
* History of tetracycline therapy within the past 6 months;
* Pregnancy or patient intending to become pregnant within the 9 months of the trial period. For women of child-bearing potential, a pregnancy test will be performed;
* Sexually active women of child-bearing potential not actively practicing birth control by using a medically accepted device or therapy (i.e., intrauterine device, hormonal contraceptive, or barrier device) during the study period (at least 24 months). This is important as doxycycline may interfere with the effectiveness of hormonal contraceptives. Hence, sexually active women of child-bearing potential who use a hormonal contraceptive will be required to use a second form of contraception to safeguard against contraceptive failure while participating in the study;
* Known allergy/intolerance to doxycycline, tetracyclines, or any ingredient in the study drug or placebo;
* Patients receiving phenytoin, barbiturates, carbamazepine, digoxin, or isotretinoin; patients with gastroparesis; patients with a history of gastrectomy, gastric bypass surgery, or otherwise deemed achlorhydric should all be excluded due to altered doxycycline pharmacokinetics and/or bioavailability;
* Patients taking strontium, acitretin, or tretinoin should excluded due to the potential for serious interactions with doxycycline;
* Patients with abnormal ALT or AST at baseline will be referred to their primary care physician for medical clearance for participation in this study.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Resolution of the persistent retinal fluid on optical coherence tomography (OCT) | 9 months
  percentage of patients with retinal fluid-free status

SECONDARY OUTCOMES:
Change in optical coherence tomography (OCT) central media thickness (CMT) | 9 months compared to baseline
  mean change in central media thickness
Change in best corrected visual acuity (BCVA) | 6 months and 9 months compared to Baseline
  mean change in logMAR / percentage of patients with a gain or loss of more than 5 ETDRS letters
Number of intravitreal injections (IVI) administered | 6 months and 9 months
  total number of anti-VEGF intravitreal injections
Inflammatory mediators matrix metalloproteinases MMP-9 and MMP-9 activity | Baseline, 6 months and 9 months
  anterior eye aqueous fluid and blood plasma

OTHER OUTCOMES:
Ocular Adverse Events | Baseline to 9 months
  intra-ocular pressure elevation ( more than 10 mmHg) requiring topical ocular hypertensive medications, endophthalmitis, retinal tear and detachment, uveitis, and thromboembolic events will be recorded
Systemic Adverse Events | Baseline to 9 months
  Allergy or hypersensitivity drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Elliott H Sohn, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics Department of Ophthalmology & Visual Sciences, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share the data with other researchers

REFERENCES:
- [Background] Wong WL, Su X, Li X, Cheung CM, Klein R, Cheng CY, Wong TY. Global prevalence of age-related macular degeneration and disease burden projection for 2020 and 2040: a systematic review and meta-analysis. Lancet Glob Health. 2014 Feb;2(2):e106-16. doi: 10.1016/S2214-109X(13)70145-1. Epub 2014 Jan 3. PMID 25104651
- [Background] Ferris FL 3rd, Fine SL, Hyman L. Age-related macular degeneration and blindness due to neovascular maculopathy. Arch Ophthalmol. 1984 Nov;102(11):1640-2. doi: 10.1001/archopht.1984.01040031330019. PMID 6208888
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Comparison of Age-related Macular Degeneration Treatments Trials (CATT) Research Group; Martin DF, Maguire MG, Fine SL, Ying GS, Jaffe GJ, Grunwald JE, Toth C, Redford M, Ferris FL 3rd. Ranibizumab and bevacizumab for treatment of neovascular age-related macular degeneration: two-year results. Ophthalmology. 2012 Jul;119(7):1388-98. doi: 10.1016/j.ophtha.2012.03.053. Epub 2012 May 1. PMID 22555112
- [Background] Heier JS, Brown DM, Chong V, Korobelnik JF, Kaiser PK, Nguyen QD, Kirchhof B, Ho A, Ogura Y, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Soo Y, Anderesi M, Groetzbach G, Sommerauer B, Sandbrink R, Simader C, Schmidt-Erfurth U; VIEW 1 and VIEW 2 Study Groups. Intravitreal aflibercept (VEGF trap-eye) in wet age-related macular degeneration. Ophthalmology. 2012 Dec;119(12):2537-48. doi: 10.1016/j.ophtha.2012.09.006. Epub 2012 Oct 17. PMID 23084240
- [Background] Arnold JJ, Campain A, Barthelmes D, Simpson JM, Guymer RH, Hunyor AP, McAllister IL, Essex RW, Morlet N, Gillies MC; Fight Retinal Blindness Study Group. Two-year outcomes of "treat and extend" intravitreal therapy for neovascular age-related macular degeneration. Ophthalmology. 2015 Jun;122(6):1212-9. doi: 10.1016/j.ophtha.2015.02.009. Epub 2015 Apr 4. PMID 25846847
- [Background] Brown DM, Regillo CD. Anti-VEGF agents in the treatment of neovascular age-related macular degeneration: applying clinical trial results to the treatment of everyday patients. Am J Ophthalmol. 2007 Oct;144(4):627-37. doi: 10.1016/j.ajo.2007.06.039. PMID 17893015
- [Background] Krebs I, Glittenberg C, Ansari-Shahrezaei S, Hagen S, Steiner I, Binder S. Non-responders to treatment with antagonists of vascular endothelial growth factor in age-related macular degeneration. Br J Ophthalmol. 2013 Nov;97(11):1443-6. doi: 10.1136/bjophthalmol-2013-303513. Epub 2013 Aug 21. PMID 23966368
- [Background] Barthelmes D, Walton R, Campain AE, Simpson JM, Arnold JJ, McAllister IL, Guymer RH, Hunyor AP, Essex RW, Morlet N, Gillies MC; Fight Retinal Blindness! Project Investigators. Outcomes of persistently active neovascular age-related macular degeneration treated with VEGF inhibitors: observational study data. Br J Ophthalmol. 2015 Mar;99(3):359-64. doi: 10.1136/bjophthalmol-2014-305514. Epub 2014 Sep 23. PMID 25249615
- [Background] Ersoy L, Ristau T, Kirchhof B, Liakopoulos S. Response to anti-VEGF therapy in patients with subretinal fluid and pigment epithelial detachment on spectral-domain optical coherence tomography. Graefes Arch Clin Exp Ophthalmol. 2014 Jun;252(6):889-97. doi: 10.1007/s00417-013-2519-9. Epub 2013 Nov 26. PMID 24271025
- [Background] Keane PA, Liakopoulos S, Ongchin SC, Heussen FM, Msutta S, Chang KT, Walsh AC, Sadda SR. Quantitative subanalysis of optical coherence tomography after treatment with ranibizumab for neovascular age-related macular degeneration. Invest Ophthalmol Vis Sci. 2008 Jul;49(7):3115-20. doi: 10.1167/iovs.08-1689. Epub 2008 Apr 11. PMID 18408176
- [Background] Forooghian F, Cukras C, Meyerle CB, Chew EY, Wong WT. Tachyphylaxis after intravitreal bevacizumab for exudative age-related macular degeneration. Retina. 2009 Jun;29(6):723-31. doi: 10.1097/IAE.0b013e3181a2c1c3. PMID 19516114
- [Background] Brown DM, Tuomi L, Shapiro H; Pier Study Group. Anatomical measures as predictors of visual outcomes in ranibizumab-treated eyes with neovascular age-related macular degeneration. Retina. 2013 Jan;33(1):23-34. doi: 10.1097/IAE.0b013e318263cedf. PMID 23073338
- [Background] van der Reis MI, La Heij EC, De Jong-Hesse Y, Ringens PJ, Hendrikse F, Schouten JS. A systematic review of the adverse events of intravitreal anti-vascular endothelial growth factor injections. Retina. 2011 Sep;31(8):1449-69. doi: 10.1097/IAE.0b013e3182278ab4. PMID 21817960
- [Background] Tozer K, Roller AB, Chong LP, Sadda S, Folk JC, Mahajan VB, Russell SR, Boldt HC, Sohn EH. Combination therapy for neovascular age-related macular degeneration refractory to anti-vascular endothelial growth factor agents. Ophthalmology. 2013 Oct;120(10):2029-34. doi: 10.1016/j.ophtha.2013.03.016. Epub 2013 May 25. PMID 23714319
- [Background] Veritti D, Sarao V, Lanzetta P. Bevacizumab and triamcinolone acetonide for choroidal neovascularization due to age-related macular degeneration unresponsive to antivascular endothelial growth factors. J Ocul Pharmacol Ther. 2013 May;29(4):437-41. doi: 10.1089/jop.2012.0173. Epub 2012 Dec 6. PMID 23215753
- [Background] Witkin AJ, Rayess N, Garg SJ, Maguire JI, Storey P, Kaiser RS, Hsu J, Vander JF, Ho AC. Alternating Bi-Weekly Intravitreal Ranibizumab and Bevacizumab for Refractory Neovascular Age-Related Macular Degeneration with Pigment Epithelial Detachment. Semin Ophthalmol. 2017;32(3):309-315. doi: 10.3109/08820538.2015.1072222. Epub 2015 Sep 4. PMID 26337539
- [Background] Sridhar J, Hsu J, Shahlaee A, Garg SJ, Spirn MJ, Fineman MS, Vander J. Topical Dorzolamide-Timolol With Intravitreous Anti-Vascular Endothelial Growth Factor for Neovascular Age-Related Macular Degeneration. JAMA Ophthalmol. 2016 Apr;134(4):437-43. doi: 10.1001/jamaophthalmol.2016.0045. PMID 26914218
- [Background] Mirshahi A, Azimi P, Abdolahi A, Mirshahi R, Abdollahian M. Oral Doxycycline Reduces the Total Number of Intraocular Bevacizumab Injections Needed to Control Neovascular Age-related Macular Degeneration. Med Hypothesis Discov Innov Ophthalmol. 2017 Summer;6(2):23-29. PMID 29367931
- [Background] Zarbin MA. Current concepts in the pathogenesis of age-related macular degeneration. Arch Ophthalmol. 2004 Apr;122(4):598-614. doi: 10.1001/archopht.122.4.598. PMID 15078679
- [Background] Ambati J, Ambati BK, Yoo SH, Ianchulev S, Adamis AP. Age-related macular degeneration: etiology, pathogenesis, and therapeutic strategies. Surv Ophthalmol. 2003 May-Jun;48(3):257-93. doi: 10.1016/s0039-6257(03)00030-4. PMID 12745003
- [Background] Schaal S, Kaplan HJ, Tezel TH. Is there tachyphylaxis to intravitreal anti-vascular endothelial growth factor pharmacotherapy in age-related macular degeneration? Ophthalmology. 2008 Dec;115(12):2199-205. doi: 10.1016/j.ophtha.2008.07.007. Epub 2008 Oct 18. PMID 18930553
- [Background] Binder S. Loss of reactivity in intravitreal anti-VEGF therapy: tachyphylaxis or tolerance? Br J Ophthalmol. 2012 Jan;96(1):1-2. doi: 10.1136/bjophthalmol-2011-301236. No abstract available. PMID 22157632
- [Background] Steen B, Sejersen S, Berglin L, Seregard S, Kvanta A. Matrix metalloproteinases and metalloproteinase inhibitors in choroidal neovascular membranes. Invest Ophthalmol Vis Sci. 1998 Oct;39(11):2194-200. PMID 9761302
- [Background] Tatar O, Adam A, Shinoda K, Eckert T, Scharioth GB, Klein M, Yoeruek E, Bartz-Schmidt KU, Grisanti S. Matrix metalloproteinases in human choroidal neovascular membranes excised following verteporfin photodynamic therapy. Br J Ophthalmol. 2007 Sep;91(9):1183-9. doi: 10.1136/bjo.2007.114769. Epub 2007 May 2. PMID 17475706
- [Background] Nussenblatt RB, Ferris F 3rd. Age-related macular degeneration and the immune response: implications for therapy. Am J Ophthalmol. 2007 Oct;144(4):618-26. doi: 10.1016/j.ajo.2007.06.025. Epub 2007 Aug 15. PMID 17698021
- [Background] Johnson LV, Anderson DH. Age-related macular degeneration and the extracellular matrix. N Engl J Med. 2004 Jul 22;351(4):320-2. doi: 10.1056/NEJMp048131. No abstract available. PMID 15269309
- [Background] Ng EW, Adamis AP. Targeting angiogenesis, the underlying disorder in neovascular age-related macular degeneration. Can J Ophthalmol. 2005 Jun;40(3):352-68. doi: 10.1016/S0008-4182(05)80078-X. PMID 15947805
- [Background] Spraul CW, Lang GE, Grossniklaus HE, Lang GK. Histologic and morphometric analysis of the choroid, Bruch's membrane, and retinal pigment epithelium in postmortem eyes with age-related macular degeneration and histologic examination of surgically excised choroidal neovascular membranes. Surv Ophthalmol. 1999 Oct;44 Suppl 1:S10-32. doi: 10.1016/s0039-6257(99)00086-7. PMID 10548114
- [Background] Chong NH, Keonin J, Luthert PJ, Frennesson CI, Weingeist DM, Wolf RL, Mullins RF, Hageman GS. Decreased thickness and integrity of the macular elastic layer of Bruch's membrane correspond to the distribution of lesions associated with age-related macular degeneration. Am J Pathol. 2005 Jan;166(1):241-51. doi: 10.1016/S0002-9440(10)62248-1. PMID 15632016
- [Background] Egeblad M, Werb Z. New functions for the matrix metalloproteinases in cancer progression. Nat Rev Cancer. 2002 Mar;2(3):161-74. doi: 10.1038/nrc745. PMID 11990853
- [Background] Overall CM, Lopez-Otin C. Strategies for MMP inhibition in cancer: innovations for the post-trial era. Nat Rev Cancer. 2002 Sep;2(9):657-72. doi: 10.1038/nrc884. PMID 12209155
- [Background] Shapiro SD. Matrix metalloproteinase degradation of extracellular matrix: biological consequences. Curr Opin Cell Biol. 1998 Oct;10(5):602-8. doi: 10.1016/s0955-0674(98)80035-5. PMID 9818170
- [Background] Lund LR, Romer J, Bugge TH, Nielsen BS, Frandsen TL, Degen JL, Stephens RW, Dano K. Functional overlap between two classes of matrix-degrading proteases in wound healing. EMBO J. 1999 Sep 1;18(17):4645-56. doi: 10.1093/emboj/18.17.4645. PMID 10469644
- [Background] Wissink S, van Heerde EC, Schmitz ML, Kalkhoven E, van der Burg B, Baeuerle PA, van der Saag PT. Distinct domains of the RelA NF-kappaB subunit are required for negative cross-talk and direct interaction with the glucocorticoid receptor. J Biol Chem. 1997 Aug 29;272(35):22278-84. doi: 10.1074/jbc.272.35.22278. PMID 9268377
- [Background] Kvanta A, Shen WY, Sarman S, Seregard S, Steen B, Rakoczy E. Matrix metalloproteinase (MMP) expression in experimental choroidal neovascularization. Curr Eye Res. 2000 Sep;21(3):684-90. PMID 11120556
- [Background] Kvanta A, Sarman S, Fagerholm P, Seregard S, Steen B. Expression of matrix metalloproteinase-2 (MMP-2) and vascular endothelial growth factor (VEGF) in inflammation-associated corneal neovascularization. Exp Eye Res. 2000 Apr;70(4):419-28. doi: 10.1006/exer.1999.0790. PMID 10865990
- [Background] Guo L, Hussain AA, Limb GA, Marshall J. Age-dependent variation in metalloproteinase activity of isolated human Bruch's membrane and choroid. Invest Ophthalmol Vis Sci. 1999 Oct;40(11):2676-82. PMID 10509665
- [Background] Kamei M, Hollyfield JG. TIMP-3 in Bruch's membrane: changes during aging and in age-related macular degeneration. Invest Ophthalmol Vis Sci. 1999 Sep;40(10):2367-75. PMID 10476804
- [Background] Fiotti N, Pedio M, Battaglia Parodi M, Altamura N, Uxa L, Guarnieri G, Giansante C, Ravalico G. MMP-9 microsatellite polymorphism and susceptibility to exudative form of age-related macular degeneration. Genet Med. 2005 Apr;7(4):272-7. doi: 10.1097/01.gim.0000159903.69597.73. PMID 15834245
- [Background] Oshima Y, Oshima S, Nambu H, Kachi S, Hackett SF, Melia M, Kaleko M, Connelly S, Esumi N, Zack DJ, Campochiaro PA. Increased expression of VEGF in retinal pigmented epithelial cells is not sufficient to cause choroidal neovascularization. J Cell Physiol. 2004 Dec;201(3):393-400. doi: 10.1002/jcp.20110. PMID 15389527
- [Background] Samtani S, Amaral J, Campos MM, Fariss RN, Becerra SP. Doxycycline-mediated inhibition of choroidal neovascularization. Invest Ophthalmol Vis Sci. 2009 Nov;50(11):5098-106. doi: 10.1167/iovs.08-3174. Epub 2009 Jun 10. PMID 19516001
- [Background] Roychoudhury J, Herndon JM, Yin J, Apte RS, Ferguson TA. Targeting immune privilege to prevent pathogenic neovascularization. Invest Ophthalmol Vis Sci. 2010 Jul;51(7):3560-6. doi: 10.1167/iovs.09-3890. Epub 2010 Feb 17. PMID 20164456
- [Background] Schwesinger C, Yee C, Rohan RM, Joussen AM, Fernandez A, Meyer TN, Poulaki V, Ma JJ, Redmond TM, Liu S, Adamis AP, D'Amato RJ. Intrachoroidal neovascularization in transgenic mice overexpressing vascular endothelial growth factor in the retinal pigment epithelium. Am J Pathol. 2001 Mar;158(3):1161-72. doi: 10.1016/S0002-9440(10)64063-1. PMID 11238064
- [Background] Ogata N, Wada M, Otsuji T, Jo N, Tombran-Tink J, Matsumura M. Expression of pigment epithelium-derived factor in normal adult rat eye and experimental choroidal neovascularization. Invest Ophthalmol Vis Sci. 2002 Apr;43(4):1168-75. PMID 11923262
- [Background] Dawson DW, Volpert OV, Gillis P, Crawford SE, Xu H, Benedict W, Bouck NP. Pigment epithelium-derived factor: a potent inhibitor of angiogenesis. Science. 1999 Jul 9;285(5425):245-8. doi: 10.1126/science.285.5425.245. PMID 10398599
- [Background] Becerra SP. Focus on Molecules: Pigment epithelium-derived factor (PEDF). Exp Eye Res. 2006 May;82(5):739-40. doi: 10.1016/j.exer.2005.10.016. Epub 2005 Dec 20. No abstract available. PMID 16364294
- [Background] Gehlbach P, Demetriades AM, Yamamoto S, Deering T, Duh EJ, Yang HS, Cingolani C, Lai H, Wei L, Campochiaro PA. Periocular injection of an adenoviral vector encoding pigment epithelium-derived factor inhibits choroidal neovascularization. Gene Ther. 2003 Apr;10(8):637-46. doi: 10.1038/sj.gt.3301931. PMID 12692592
- [Background] Lambert V, Munaut C, Jost M, Noel A, Werb Z, Foidart JM, Rakic JM. Matrix metalloproteinase-9 contributes to choroidal neovascularization. Am J Pathol. 2002 Oct;161(4):1247-53. doi: 10.1016/S0002-9440(10)64401-X. PMID 12368198
- [Background] Lambert V, Wielockx B, Munaut C, Galopin C, Jost M, Itoh T, Werb Z, Baker A, Libert C, Krell HW, Foidart JM, Noel A, Rakic JM. MMP-2 and MMP-9 synergize in promoting choroidal neovascularization. FASEB J. 2003 Dec;17(15):2290-2. doi: 10.1096/fj.03-0113fje. Epub 2003 Oct 16. PMID 14563686
- [Background] Bergers G, Brekken R, McMahon G, Vu TH, Itoh T, Tamaki K, Tanzawa K, Thorpe P, Itohara S, Werb Z, Hanahan D. Matrix metalloproteinase-9 triggers the angiogenic switch during carcinogenesis. Nat Cell Biol. 2000 Oct;2(10):737-44. doi: 10.1038/35036374. PMID 11025665
- [Background] Hollborn M, Stathopoulos C, Steffen A, Wiedemann P, Kohen L, Bringmann A. Positive feedback regulation between MMP-9 and VEGF in human RPE cells. Invest Ophthalmol Vis Sci. 2007 Sep;48(9):4360-7. doi: 10.1167/iovs.06-1234. PMID 17724228
- [Background] Liutkeviciene R, Lesauskaite V, Sinkunaite-Marsalkiene G, Zaliuniene D, Zaliaduonyte-Peksiene D, Mizariene V, Gustiene O, Jasinskas V, Jariene G, Tamosiunas A. The Role of Matrix Metalloproteinases Polymorphisms in Age-Related Macular Degeneration. Ophthalmic Genet. 2015 Jun;36(2):149-55. doi: 10.3109/13816810.2013.838274. Epub 2013 Sep 30. PMID 24079541
- [Background] Chau KY, Sivaprasad S, Patel N, Donaldson TA, Luthert PJ, Chong NV. Plasma levels of matrix metalloproteinase-2 and -9 (MMP-2 and MMP-9) in age-related macular degeneration. Eye (Lond). 2008 Jun;22(6):855-9. PMID 18597988
- [Background] Jonas JB, Tao Y, Neumaier M, Findeisen P. Cytokine concentration in aqueous humour of eyes with exudative age-related macular degeneration. Acta Ophthalmol. 2012 Aug;90(5):e381-8. doi: 10.1111/j.1755-3768.2012.02414.x. Epub 2012 Apr 10. PMID 22490043
- [Background] Thode AR, Latkany RA. Current and Emerging Therapeutic Strategies for the Treatment of Meibomian Gland Dysfunction (MGD). Drugs. 2015 Jul;75(11):1177-85. doi: 10.1007/s40265-015-0432-8. PMID 26130187
- [Background] Ochsendorf F. Systemic antibiotic therapy of acne vulgaris. J Dtsch Dermatol Ges. 2006 Oct;4(10):828-41. doi: 10.1111/j.1610-0387.2006.06053.x. English, German. PMID 17010172
- [Background] Cunha BA. New uses for older antibiotics: nitrofurantoin, amikacin, colistin, polymyxin B, doxycycline, and minocycline revisited. Med Clin North Am. 2006 Nov;90(6):1089-107. doi: 10.1016/j.mcna.2006.07.006. PMID 17116438
- [Background] Doughty MJ. On the prescribing of oral doxycycline or minocycline by UK optometrists as part of management of chronic Meibomian Gland Dysfunction (MGD). Cont Lens Anterior Eye. 2016 Feb;39(1):2-8. doi: 10.1016/j.clae.2015.08.002. Epub 2015 Sep 4. PMID 26347083
- [Background] Burns FR, Stack MS, Gray RD, Paterson CA. Inhibition of purified collagenase from alkali-burned rabbit corneas. Invest Ophthalmol Vis Sci. 1989 Jul;30(7):1569-75. PMID 2545645
- [Background] Golub LM, Sorsa T, Lee HM, Ciancio S, Sorbi D, Ramamurthy NS, Gruber B, Salo T, Konttinen YT. Doxycycline inhibits neutrophil (PMN)-type matrix metalloproteinases in human adult periodontitis gingiva. J Clin Periodontol. 1995 Feb;22(2):100-9. doi: 10.1111/j.1600-051x.1995.tb00120.x. PMID 7775665
- [Background] Golub LM, Lee HM, Ryan ME, Giannobile WV, Payne J, Sorsa T. Tetracyclines inhibit connective tissue breakdown by multiple non-antimicrobial mechanisms. Adv Dent Res. 1998 Nov;12(2):12-26. doi: 10.1177/08959374980120010501. PMID 9972117
- [Background] Sorsa T, Ding Y, Salo T, Lauhio A, Teronen O, Ingman T, Ohtani H, Andoh N, Takeha S, Konttinen YT. Effects of tetracyclines on neutrophil, gingival, and salivary collagenases. A functional and western-blot assessment with special reference to their cellular sources in periodontal diseases. Ann N Y Acad Sci. 1994 Sep 6;732:112-31. doi: 10.1111/j.1749-6632.1994.tb24729.x. PMID 7978785
- [Background] Garcia RA, Pantazatos DP, Gessner CR, Go KV, Woods VL Jr, Villarreal FJ. Molecular interactions between matrilysin and the matrix metalloproteinase inhibitor doxycycline investigated by deuterium exchange mass spectrometry. Mol Pharmacol. 2005 Apr;67(4):1128-36. doi: 10.1124/mol.104.006346. Epub 2005 Jan 21. PMID 15665254
- [Background] Alvarenga LS, Mannis MJ. Ocular rosacea. Ocul Surf. 2005 Jan;3(1):41-58. doi: 10.1016/s1542-0124(12)70121-0. PMID 17131004
- [Background] Notari L, Miller A, Martinez A, Amaral J, Ju M, Robinson G, Smith LE, Becerra SP. Pigment epithelium-derived factor is a substrate for matrix metalloproteinase type 2 and type 9: implications for downregulation in hypoxia. Invest Ophthalmol Vis Sci. 2005 Aug;46(8):2736-47. doi: 10.1167/iovs.04-1489. PMID 16043845
- [Background] Barber AJ, Gardner TW, Abcouwer SF. The significance of vascular and neural apoptosis to the pathology of diabetic retinopathy. Invest Ophthalmol Vis Sci. 2011 Feb 28;52(2):1156-63. doi: 10.1167/iovs.10-6293. Print 2011 Feb. PMID 21357409
- [Background] Scott IU, Jackson GR, Quillen DA, Klein R, Liao J, Gardner TW. Effect of doxycycline vs placebo on retinal function and diabetic retinopathy progression in mild to moderate nonproliferative diabetic retinopathy: a randomized proof-of-concept clinical trial. JAMA Ophthalmol. 2014 Sep;132(9):1137-42. doi: 10.1001/jamaophthalmol.2014.1422. PMID 24969516